CLINICAL TRIAL: NCT07233759
Title: The Theraprutic Effect of New Drugs for Hepatocellular Carcinoma
Brief Title: The Study Collect Clinical Data From the Treatment of Liver Cancer With New Drugs After 2019 and Integrate Biochemical and Pathological Indicators to Analyze Prognostic Outcomes, Including Overall Survival, Progression-free Survival, and Complications.
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202212042RINA
Record Dates: First submitted 2025-10-01; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Liver Cancer; Pembrolizumab; Atezolizumab; Lenvatinib
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most significant cancers in our country. Since 2019, many first-line and second-line therapeutic agents for HCC have been introduced. This study aims to evaluate the treatment outcomes of HCC patients in our hospital from 2019 to 2024 who received therapies other than the traditional sorafenib (Nexavar). The included drugs are Pembrolizumab, Atezolizumab (Tecentriq), Nivolumab, Lenvatinib, and Regorafenib (Stivarga). The study will collect clinical data from treated-cases with these novel agents after 2019 and integrate biochemical and pathological indicators to analyze prognostic outcomes, including overall survival, progression-free survival, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma participants who received treatment at National Taiwan University Hospital between January 1, 2019, and June 30, 2026, and had used the following medications.

  1. Pembrolizumab /keytruda
  2. Atezolizumab / Tecentriq
  3. Nivolumab
  4. Lenvatinib
  5. Stivarga

     Exclusion Criteria:
* None

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma participants who received treatment
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
liver cancer response of evaluation according to RECIST and mRECIST criteria | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided